CLINICAL TRIAL: NCT04759755
Title: Circadian and Sleep Pathways to Cardiometabolic Disease Risk: Role of Neurobehavioral Processes
Brief Title: Circadian Timing, Information Processing and Energy Balance Study
Acronym: TIME
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Rush University Medical Center (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kelly Glazer Baron, Associate Professor, University of Utah
Other Study IDs: 00117438; 1R01HL141706-01A1 (NIH)
Record Dates: First submitted 2021-02-13; First posted 2021-02-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: None Retained — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: 18-60 year olds who demonstrate habitual sleep onset time between 10:00 pm-3:00 am and BMI 25-39.9.

SUMMARY:
This study design will test biological and behavioral mechanisms in the cross-sectional analyses and determine the prospective effects of circadian alignment and sleep on changes in cardiometabolic risk factors.

DETAILED DESCRIPTION:
The goal of this study is to determine how sleep and circadian rhythm alignment contribute to neurobehavioral and behavioral mechanisms of cardiometabolic risk. The investigators propose that circadian misalignment, which is more common among individuals with late sleep timing, leads to increased consumption of energy dense/prepared foods and to decreased insulin sensitivity. Short sleep duration and neurobehavioral measures (i.e. delay discounting) may moderate these associations, thus exacerbating cardiometabolic risk factors. There is evidence for a direct biological link between circadian misalignment and insulin resistance, and for a relationship that is mediated through changes in eating behaviors. Insulin resistance and increased caloric intake over time lead to increased BMI and body fat.

In this study, the investigators will conduct cross-sectional and longitudinal analyses to determine biological and behavioral mechanisms that link circadian alignment and sleep duration to changes in cardiometabolic risk over 1 year. This study will identify individual differences that predict risk for cardiometabolic disorders and suggest potential for sleep, circadian and neurobehavioral interventions to reduce cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate habitual sleep onset time between 10:00 pm-3:00 am on actigraphy;
* able to read and write in English;
* BMI 25-39.9 (overweight, class one obesity, or class two obesity)

Exclusion Criteria:

* High risk or presence of sleep disorders (obstructive sleep apnea (OSA), restless legs syndrome, or insomnia) as assessed by the questionnaires and overnight OSA screening;
* Diagnosed with diabetes or HbA1c>7 at screening or taking medications known to affect glucose;
* History of cognitive or neurological disorders;
* Presence of major psychiatric disorders, current alcohol or substance abuse as determined by screening questionnaires or self-report;
* Unstable or serious medical illness;
* Overnight shift work or travel over 2 time zones in the past 2 months;
* Use of hypnotic, stimulant or medications know to affect melatonin concentrations such as beta blockers, daily NSAIDs;
* Current smoking;
* Daily caffeine intake >300 mg;
* Pregnant or lactating;
* Currently on a restrictive of special diet.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | Baseline
  Measured by a frequently sampled IV glucose tolerance test

SECONDARY OUTCOMES:
Eating behaviors | 12 months
  Healthy Eating Index will be calculated from the Automated Self-Assessment of 24 hour diet recall (ASA-24)
Delay discounting | Baseline
  Measured by a 10 item adjusting delay discounting measure

OTHER OUTCOMES:
Body mass index | 12 months
  Height and weight will be measured at screening and 1 year follow-up
Metabolic control | 12 months
  HbA1c will be measured at screening and 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request
Time Frame: Data will be available within 1 year of completion of the study and will be available for 1 year
Access Criteria: Written request to the PI

REFERENCES:
- [Derived] Baron KG, Appelhans BM, Burgess HJ, Quinn L, Greene T, Allen CM. Circadian Timing, Information processing and Metabolism (TIME) study: protocol of a longitudinal study of sleep duration, circadian alignment and cardiometabolic health among overweight adults. BMC Endocr Disord. 2023 Jan 31;23(1):26. doi: 10.1186/s12902-023-01272-y. PMID 36717911